CLINICAL TRIAL: NCT01199965
Title: An Open-Label, 2-Period, Crossover Phase 2 Study Comparing the Pharmacokinetics and Tolerability of Dihydroergotamine Mesylate (DHE) Delivered Intravenously (DHE 45) and by Oral Inhalation (MAP0004) in Smoking and Non-Smoking Adult Volunteers
Brief Title: Pharmacokinetics & Tolerability Study of MAP0004 in Smoking and Non-Smoking Adult Volunteers
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Allergan (Industry)
Collaborators: MAP Pharmaceuticals, Inc., a wholly owned subsidiary of Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MAP0004-CL-P203
Record Dates: First submitted 2010-08-05; First posted 2010-09-13 (Estimated); Results first posted 2013-10-22 (Estimated); Last update posted 2014-01-09 (Estimated); Status verified 2013-12

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — Dihydroergotamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IV DHE then MAP0004 (Other): Smokers and non-smokers received Intravenous Dihydroergotamine Mesylate (IV DHE) at Visit 2 followed by MAP0004 7-11 days later at Visit 3.
  Interventions: Drug: MAP0004; Drug: IV DHE
- MAP0004 then IV DHE (Other): Smokers and non-smokers received MAP0004 at Visit 2 followed by Intravenous Dihydroergotamine Mesylate (IV DHE) 7-11 days later at Visit 3.
  Interventions: Drug: MAP0004; Drug: IV DHE

INTERVENTIONS:
Drug: MAP0004 — 1.0mg MAP0004 via inhalation at Visit 2 or 3 as per protocol
Drug: IV DHE — IV DHE administered at Visit 2 or 3 as per protocol
  Other Names: D.H.E.45®

SUMMARY:
Compare the pharmacokinetics of Dihydroergotamine Mesylate (DHE) delivered by oral inhalation (MAP0004) or Intravenous (IV) DHE in smokers versus non-smokers.

Identify whether there are clinically significant differences in the tolerability of MAP0004 between smokers and non-smokers.

ELIGIBILITY:
Major Inclusion Criteria:

1. Able to provide written informed consent
2. Male or Female subjects 18 to 45 years old
3. Female subjects who are practicing adequate contraception or who are sterile
4. Stable cardiac status
5. Normal rhythm or arrhythmia deemed clinically insignificant on ECG

Major Exclusion Criteria:

1. Contraindication to dihydroergotamine mesylate (DHE)
2. Use of any excluded concomitant medications within the 10 days prior to Visit 1 (See Section 5.5)
3. History of hemiplegic or basilar migraine
4. Participation in another investigational trial during the 30 days prior to Visit 1 or during this trial

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2010-01; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Simbec Research Limited, Merthyr Tydfil, Merthyr Tydfil, United Kingdom

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All smoking and non-smoking subjects received both MAP0004 and Intravenous (IV) Dihydroergotamine (DHE).
Groups:
- Smokers: Currently smoking at least 10 cigarettes/day for at least 1 year with a positive urinary cotinine result.
- Non-smokers: Never smoked or total exposure <1 pack year and at least 12 months since last cigarette with a negative urinary cotinine result at screening.
Period: Overall Study
Arm/Group | Smokers | Non-smokers
Started | 23 | 24
Completed | 22 | 24
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Smokers | Non-smokers | Total
Number analyzed (Participants) | 23 | 24 | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.91 (7.1) | 30.71 (8.8) | 31.79 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 16 | 31
  Male | 8 | 8 | 16

OUTCOME MEASURES:

1. Primary Outcome: Cmax of Dihydroergotamine After MAP0004 and IV DHE Administration in Smokers Versus Non-smokers
Description: The maximum concentration (Cmax) is the highest concentration of a drug measured in the plasma. Plasma is the clear portion of the blood. The Cmax of Dihydroergotamine is reported in picograms per milliliter (pg/ml).
Time Frame: 48 hours
Population: Patients with available data at specified time points are included in the analysis population.
Measure: Geometric Mean (Standard Deviation); unit: pg/ml
Groups:
- MAP0004 1.0mg Smokers: Currently smoking at least 10 cigarettes/day for at least 1 year with a positive urinary cotinine result and receiving MAP0004 at either Visit 2 or 3.
- MAP0004 1.0mg Non-smokers: Never smoked or total exposure <1 pack year and at least 12 months since last cigarette with a negative urinary cotinine result at screening and receiving MAP0004 at either Visit 2 or 3.
- IV DHE 1.0mg Smokers: Currently smoking at least 10 cigarettes/day for at least 1 year with a positive urinary cotinine result and receiving IV DHE at either Visit 2 or 3.
- IV DHE 1.0mg Non-smokers: Never smoked or total exposure <1 pack year and at least 12 months since last cigarette with a negative urinary cotinine result at screening and receiving IV DHE at either Visit 2 or 3.
Arm/Group | MAP0004 1.0mg Smokers | MAP0004 1.0mg Non-smokers | IV DHE 1.0mg Smokers | IV DHE 1.0mg Non-smokers
Number analyzed (Participants) | 22 | 24 | 22 | 24
pg/ml | 1282.059 (636.138) | 2550.727 (1297.097) | 60046.128 (49580.385) | 48428.635 (43894.253)

2. Primary Outcome: AUC(0-48) of Dihydroergotamine After MAP0004 and IV DHE Administration in Smokers and Non-smokers
Description: The AUC(0-48) is the area under the plot of plasma concentration of drug against time after drug administration. Dihydroergotamine AUC(0-48) is reported in picograms times hour per milliliter (pg*h/ml).
Time Frame: 48 hours
Population: Patients with available data at specified time points are included in the analysis population.
Measure: Geometric Mean (Standard Deviation); unit: pg*h/ml
Groups:
- MAP0004 1.0mg Smokers: Currently smoking at least 10 cigarettes/day for at least 1 year with a positive urinary cotinine result and receiving MAP0004 at Visit 2 or 3.
- MAP0004 1.0mg Non-smokers: Never smoked or total exposure <1 pack year and at least 12 months since last cigarette with a negative urinary cotinine result at screening and receiving MAP0004 at Visit 2 or 3.
- IV DHE 1.0mg Smokers: Currently smoking at least 10 cigarettes/day for at least 1 year with a positive urinary cotinine result and receiving IV DHE at Visit 2 or 3.
- IV DHE 1.0mg Non-smokers: Never smoked or total exposure <1 pack year and at least 12 months since last cigarette with a negative urinary cotinine result at screening and receiving IV DHE at Visit 2 or 3.
Arm/Group | MAP0004 1.0mg Smokers | MAP0004 1.0mg Non-smokers | IV DHE 1.0mg Smokers | IV DHE 1.0mg Non-smokers
Number analyzed (Participants) | 23 | 24 | 22 | 24
pg*h/ml | 3014.968 (1136.162) | 4148.750 (1533.861) | 11049.027 (3744.094) | 11731.639 (3167.828)

ADVERSE EVENTS:
Description: All 24 non-smoking subjects who received MAP0004 and IV DHE and 23 smoking subjects who received MAP0004 and 22 of the 23 smoking subjects received IV DHE were included in the adverse event analysis.
Arm/Group | MAP0004 1.0mg Smokers | MAP0004 1.0mg Non-smokers | IV DHE 1.0mg Smokers | IV DHE 1.0mg Non-smokers
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/24 | 0/22 | 0/24
Other Adverse Events (participants affected / at risk) | 4/23 | 8/24 | 15/22 | 22/24
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MAP0004 1.0mg Smokers (N=23) | MAP0004 1.0mg Non-smokers (N=24) | IV DHE 1.0mg Smokers (N=22) | IV DHE 1.0mg Non-smokers (N=24)
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 2
Dizziness (Nervous system disorders) | 1 | 1 | 6 | 2
Headache (Nervous system disorders) | 2 | 2 | 6 | 10
Paraesthesia (Nervous system disorders) | 0 | 2 | 1 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Flushing (Vascular disorders) | 0 | 0 | 2 | 5
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 2
Nausea (Gastrointestinal disorders) | 1 | 0 | 5 | 9
Vomiting (Gastrointestinal disorders) | 0 | 0 | 2 | 5
Rhinitis (Infections and infestations) | 0 | 2 | 0 | 1
Chest discomfort (General disorders) | 0 | 0 | 2 | 3
Fatigue (General disorders) | 0 | 1 | 2 | 0
Feeling hot (General disorders) | 0 | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.